CLINICAL TRIAL: NCT03644693
Title: Evaluation of the Safety and Tolerability of a Nutritional Formulation in Angelman Syndrome
Brief Title: Nutritional Formulation for Angelman Syndrome
Acronym: FANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 20-0366
Record Dates: First submitted 2018-08-13; First posted 2018-08-23 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome; Ketosis; Children
MeSH Terms: conditions — Angelman Syndrome; Ketosis

STUDY DESIGN:
Intervention Model Description: The study design for this nutritional intervention protocol is a randomized, double blind, placebo controlled crossover study. Each patient will receive both nutritional formulation and placebo formulation, with a washout period between each arm. The dietary backgrounds will differ among patients. Acceptable diets include three basic diets: ketogenic diet (i.e. conventional 4:1 or 3:1, modified Atkins), low glycemic index diet (LGIT), and standard American diet (regular diet).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): Subjects assigned to this arm will receive the Nutritional Formulation containing exogenous ketones.
  Interventions: Dietary Supplement: Nutritional Formulation Containing Exogenous Ketones
- Placebo (Placebo Comparator): Subjects assigned to this arm will receive the Placebo Formulation.
  Interventions: Dietary Supplement: Placebo Formulation

INTERVENTIONS:
Dietary Supplement: Nutritional Formulation Containing Exogenous Ketones — A nutritional formulation providing beta-hydroxybutyrate, 2g of carbohydrate, 1g of protein, and 9g of fat, plus minerals, per 100kcal. Given orally as food or beverage three times daily.
  Arms: Investigational
Dietary Supplement: Placebo Formulation — A placebo formulation providing similar amounts of carbohydrates, proteins and minerals as the nutritional formulation. Given orally as food or beverage three times daily.
  Arms: Placebo

SUMMARY:
Low carbohydrate diets such as the ketogenic (KD) and low glycemic index (LGIT) diets have been shown to be effective in treating drug resistant seizures in children with Angelman syndrome (AS). The investigators hypothesize that consuming a fat based nutritional formulation with an exogenous ketone throughout the day will produce urinary ketosis in children consuming both low and high carbohydrate diets, depending upon dietary background. The nutritional formulation will provide fuel substrates that push metabolism away from carbohydrates and towards fat utilization. This research is being done to assess the safety and tolerability of a nutritional formulation for use in dietary interventions in AS.

DETAILED DESCRIPTION:
An evaluation of the safety and tolerability of a nutritional formulation in Angelman syndrome in children ages 4-11 years.

Study is conducted over 16 weeks:

2 week baseline period - Patient continues on current dietary regimen they were on before joining the study (standard, ketogenic, or LGIT).

4 week intervention period - Patient consumes either placebo or nutritional formulation for 4 weeks, maintaining their current diet.

4 week washout period - Patient continues on current dietary regimen without consuming any study formulations.

4 week intervention period - Patient consumes either placebo or nutritional formulation for 4 weeks (crossover), maintaining their current diet.

2 week washout period - Patient continues on current dietary regimen without consuming any study formulations.

Follow-up phone call to be conducted by study personnel during this time.

Data is captured by the investigator during baseline, intervention, and washout periods, and by the parent/caregiver daily throughout the protocol using apps loaded on a provided tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 4-11 years of age
* Diagnosed with Angelman syndrome with prior lab report indicating genetic diagnosis
* Currently on a LGIT, KD, or standard diet consistently for at least three months
* Motivated to maintain the LGIT or KD for at least the duration of the trial period, as applicable
* Written informed consent from patient and/or parent/caregiver
* Willing to drink provided formulations, or to eat them mixed with food
* Daytime toilet trained, or parents willing to use cotton balls in diapers to sample urine
* Willing to test urine daily
* Willing to comply with protocol examinations, including EEG, ERP, and venipuncture
* Ambulatory, willing to perform gait tracking

Exclusion Criteria:

* Being pregnant or planning pregnancy
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* History of a diagnosis of diabetes
* Participation in other clinical intervention studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients
* Investigator concern around willingness/ability of patient or parent/caregiver to comply with protocol requirements
* Any contraindications for the use of the ketogenic or low carbohydrate diets
* Significantly underweight (Body Mass Index <18.5)
* Unwilling to drink provided formulations, or to consume formulation mixed with food
* Not ambulatory, or unwilling to perform gait tracking
* Not daytime toilet trained, or parents unwilling to use cotton balls in diapers to sample urine
* Unwilling to test urine daily

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Compliance with feeding protocol | 16 weeks
  Tolerability will be demonstrated through patient compliance with the protocol as determined by the amount as measured in grams per day of nutritional formulation consumed as compared to the amount prescribed.

SECONDARY OUTCOMES:
Convenience, taste, and acceptability | 16 weeks (measured 2 times)
  Parents/caregivers will rate convenience, taste, and acceptability of the nutritional formulation on a ten-point Likert scale. Each parameter will be rated individually with 1 = poor and 10 = excellent.
Urinary Ketosis | 16 weeks
  The degree of nutritional ketosis will be evaluated in patients with different dietary backgrounds when consuming the nutritional formulation. Urine ketones will be recorded daily as mmol of acetoacetate.
Serum Ketosis | 16 weeks (measured 3 times)
  The degree of nutritional ketosis will be evaluated in patients with different dietary backgrounds when consuming the nutritional formulation. Serum ketones will be recorded as mmol of R-beta-hydroxybutyrate.
Number of Patients with Adverse Events | 16 weeks (measured 3 times)
  All adverse events will be monitored throughout the study. The number and type of adverse event will be recorded.
Change in Mobility Measured Using Zeno Walkway | 16 weeks (measured 3 times)
  Patients with Angelman Syndrome typically have motor coordination and physical developmental delays resulting in an ataxic gate. As a measure of safety, the patient's gate characteristics for cadence will be compared to baseline.
Change in Cognition as Measured by Event Related Potentials (ERP) | 16 weeks (measured 3 times)
  Patients with Angelman Syndrome have global severe intellectual disability. As a measure of safety, ERP waveform amplitude and timing in response to a presented stimuli will be compared to baseline.
Change in Cortical Irritability Measured Using Electroencephalogram (EEG) | 16 weeks (measured 3 times)
  Patients with Angelman Syndrome have a characteristic EEG signature and are prone to seizure. As a measure of safety, the EEG signature will be compared to baseline in terms of the numbers of epileptiform discharges, notched delta and rhythmic theta activity.
Number of Patients with Treatment Related Adverse Events as Assessed by Blood Metabolic Panel | 16 weeks (measured 3 times)
  Blood samples will be taken and assessed for complete blood count, comprehensive metabolic panel, ketones, and lipids.
Nutrient Intake | 16 weeks
  Food diaries recorded daily to establish total caloric and macro-nutrient intake.
Changes in Gastrointestinal (GI) Health | 16 weeks
  Patients with Angelman Syndrome frequently suffer from poor GI health. As a measure of safety, bowel movements will be characterized daily according to the Bristol Stool Chart and compared to baseline.
Changes in Sleep | 16 weeks
  Patients with Angelman Syndrome frequently suffer from sleep issues. As a measure of safety, sleep duration and stage will be characterized by recording movement, heart rate and breathing during nighttime sleep and compared to baseline.
Changes in Seizures | 16 weeks
  A significant percentage of Patients with Angelman Syndrome suffer from epileptic seizures. As a measure of safety, the number and type of seizures that occur will be recorded daily in a diary and compare to baseline.
Height | 16 weeks (measured 3 times)
  Height (cm)
Weight | 16 weeks (measured 3 times)
  Weight (kg)
Change from Baseline in the Vineland Adaptive Behavior Score | 16 weeks (measured 3 times)
  Patients with Angelman Syndrome have severe global developmental delays. As a measure of safety, the Vineland Adaptive Behavior Scale, Third Edition will be used to measure changes from baseline in skills and independence.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Duis, MD, MS, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hopsital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Carson RP, Herber DL, Pan Z, Phibbs F, Key AP, Gouelle A, Ergish P, Armour EA, Patel S, Duis J. Nutritional Formulation for Patients with Angelman Syndrome: A Randomized, Double-Blind, Placebo-Controlled Study of Exogenous Ketones. J Nutr. 2021 Dec 3;151(12):3628-3636. doi: 10.1093/jn/nxab284. PMID 34510212
- [Derived] Herber DL, Weeber EJ, D'Agostino DP, Duis J. Evaluation of the safety and tolerability of a nutritional Formulation in patients with ANgelman Syndrome (FANS): study protocol for a randomized controlled trial. Trials. 2020 Jan 9;21(1):60. doi: 10.1186/s13063-019-3996-x. PMID 31918761